CLINICAL TRIAL: NCT01316315
Title: A Double-Blind, Randomized, Placebo-Controlled, Two-Period, Cross-Over Study to Evaluate the Bronchoprotective Effects of a Single Dose of N6022 in Patients With Mild Asthma
Brief Title: Study to Evaluate the Bronchoprotective Effects of a Single Dose of N6022 in Patients With Mild Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N6022-2A1-02
Record Dates: First submitted 2011-03-07; First posted 2011-03-16 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Exercise; N6022

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): N6022 - 5 mg
  Interventions: Drug: Active
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active — A 5 mg single dose given intravenously via syringe pump over 1 minute.
  Other Names: N6022
  Arms: Active
Drug: Placebo — Same as active
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a single IV dose of N6022 will have a significant bronchoprotective effect, compared with placebo, during methacholine challenge.

DETAILED DESCRIPTION:
The number of patients with adverse events measured in both the treated and placebo groups from start of dosing until Day 28 post dose.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 35 kg/m2, inclusive, at screening.
* Patient has a ≤ 5 pack years smoking history and nonsmoking for ≥ one year.
* Documented history of mild bronchial asthma, first diagnosed at least 6 months and currently being treated only with intermittent short-acting beta-agonist therapy by inhalation.
* Pre-bronchodilator FEV1 ≥ 75% of predicted at screening.
* Sensitivity to methacholine with a provocation concentration of methacholine resulting in a 20% fall in FEV1 (PC20 methacholine) of ≤ 8 mg/ml at screening.
* Demonstrated stable lung function during screening with ≤10% variability between two assessments of FEV1 taken at least 7 days apart at approximately the same time of day.

Exclusion Criteria:

* Hypertension at screening is defined as systolic blood pressure (BP) >150 mmHg or diastolic BP > 90mmHg.
* Respiratory tract infection and/or exacerbation of asthma within prior 4 weeks
* History of life-threatening asthma
* Administration of steroids within 4 weeks of the screening visit.
* History of being unable to tolerate or complete MCh testing.
* Blood donation (500 mL) within 3 months of starting the clinical study.
* Tested positive for hepatitis C antibody or hepatitis B surface antigen.
* Tested positive for human immunodeficiency virus (HIV) antibodies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhohit K Katial, MD, Principal Investigator — National Jewish Health; Monica Kraft, MD, Principal Investigator — Duke Asthma, Allergy and Airway Center
Locations (2):
- United States (2):
  - National Jewish Health, Denver, Colorado
  - Duke Asthma, Allergy and Airway Center, Durham, North Carolina

REFERENCES:
- [Derived] Que LG, Yang Z, Lugogo NL, Katial RK, Shoemaker SA, Troha JM, Rodman DM, Tighe RM, Kraft M. Effect of the S-nitrosoglutathione reductase inhibitor N6022 on bronchial hyperreactivity in asthma. Immun Inflamm Dis. 2018 Jun;6(2):322-331. doi: 10.1002/iid3.220. Epub 2018 Apr 11. PMID 29642282
- See also: Sponsor — http://n30pharma.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: N6022 - Active 5 mg
- Placebo: Non-Active
Period: Sequence 1
Arm/Group | Active | Placebo
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Sequence 2
Arm/Group | Active | Placebo
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Any patient that received a dose of N6022 or Placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Any patient that received a dose of N6022 or placebo
  Participants
    Female | 1 | 1 | 2
    Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Change in Methacholine PC20 From Baseline Compared With Placebo 24 Hours After Dosing
Description: These assessments will be recorded at various times over the study - Methacholine PC20 at screening, and at 8, 24, 48 hours postdose and Day 7; spirometry assessments will be recorded at screening, at 2, 4, 6, 8, 24, 48 hours postdose and Day 7.
Time Frame: 24 hours
Population: Any patient that received a dose of N6022 or placebo.
Measure: Mean (Standard Error); unit: mg/mL
Groups:
- N6022: Patients received a single IV administration of 5 mL of N6022 on Day 1 in each treatment period and single dose of placebo on Day 1 of the second period.
- Placebo: Patients received a single IV administration of 5 mL of placebo on Day 1 in each treatment period and single dose of N6022 on the day 1 of the second period.
Arm/Group | N6022 | Placebo
Number analyzed (Participants) | 14 | 13
mg/mL | 1.48 (.093) | -0.2 (0.3)

2. Secondary Outcome: Measurement of Change in Methacholine PC20 From Baseline Compared With Placebo 8 Hours After Dosing
Description: as for outcome 1
Time Frame: 8 hours
Population: Any patient that received a dose of N6022 or Placebo
Measure: Mean (Standard Error); unit: mg/mL
Arm/Group | Active | Placebo
Number analyzed (Participants) | 14 | 13
mg/mL | 0.3 (0.63) | -0.54 (0.33)

3. Secondary Outcome: To Assess the Safety and Tolerability of Single Dose Administration of N6022 in Patients With Mild Asthma.
Description: Adverse event (AE) reporting will begin upon signing of the consent and will continue until end-of-study (follow up phone call Day 28 +/- 2 days after dosing in the second treatment period). Number of patients with an adverse event will be documented and analyzed.
Time Frame: 10 Weeks
Population: Any patient that received a dose of N6022 or placebo
Measure: Number; unit: Adverse Events
Arm/Group | Active | Placebo
Number analyzed (Participants) | 7 | 6
Adverse Events | 11 | 9

4. Other Pre Specified Outcome: Measurement of Change in Methacholine PC20 From Baseline Compared With Placebo After 7 Days of Dosing
Time Frame: 7 Days
Population: Any patient that received a dose of N6022 or Placebo
Measure: Mean (Standard Error); unit: mg/mL
Arm/Group | Active | Placebo
Number analyzed (Participants) | 14 | 13
mg/mL | 0.74 (1.01) | -0.38 (.68)

ADVERSE EVENTS:
Time Frame: 8 Months
Description: Patients were followed from signing consent through both sequences of the crossover design.
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 11/14 | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=14) | Placebo (N=13)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection Site Hematoma (General disorders) | 2 (2) | 0 (0) — administration and site conditions
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood LDH (Investigations) | 1 (1) | 1 (1)
Blood Phosphorous Decreased (Investigations) | 2 (2) | 2 (2)
Blood Urine Present (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Turminate Abnormality (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal Erthyma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Fatigue (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic Rhinnitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erthyma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection Site Erthyma (General disorders) | 0 (0) | 1 (1) — administration and site conditions
Injection Site Induration (General disorders) | 0 (0) | 1 (1) — administration and site conditions
Injection Site Pain (General disorders) | 0 (0) | 1 (1) — administration and site conditions
Tenderness (General disorders) | 0 (0) | 3 (3) — administration and site conditions
ALT Increased (Investigations) | 1 (1) | 1 (1)
AST Increased (Investigations) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees with the use of results of the clinical study for the purposes of national and international registration, publication, and information for medical and pharmaceutical professionals. If necessary, the competent authorities will be notified of the investigator's name, address, qualifications, and extent of involvement. An investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted with the Sponsor in advance.